CLINICAL TRIAL: NCT05769803
Title: Viral Load Analysis of the SARS-CoV-2 Virus in Nose Versus Mouth Sites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-04
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Sars-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Nasal and mouth swab — Whinin 7 days from diagnosis, the subjects will be requested to sample another two specimens i.e. nasal swab and mouth swab, that will be tested for the presence of SARS-CoV-2 RNA. Results, expressed as cycle threshold will be then compared to analyze viral loads from the two different sites.
  Moreover, an aliquot will be retro-transcribed into cDNA and sequenced by Next Generation Sequencing (NGS) to obtain the virus entire genome sequence or evaluated by RT-PCR for variantdetermination.

SUMMARY:
It is a single-center, non-profit experimental study, intended to evaluate the viral load of SARS COV 2 in nasal and oral samples of positive subjects to evaluate any variation and understand which is the most suitable site for carrying out the swab.

DETAILED DESCRIPTION:
Experimental study on de-identified, biological samples (nasal and buccal swab).

The study will be performed on patients admitted to IRCCS Sacro Cuore Don Calabria Hospital or health care workers or their family members, who tested positive for SARS-CoV-2 by either a molecular or antigen test, performed on nasopharyngeal swab, according to current diagnostics.

Among the family members, also children >4 years old will be included. The reason for including children and young subjects is based on data indicating that they seems to be highly sensitive to Omicron infection and that their vaccination status could influence viral load. The nose and mouth swab are poor invasive and they could be well tolerated also by children.

Whinin 7 days from diagnosis, the subjects will be requested to sample another two specimens i.e. nasal swab and mouth swab, that will be tested for the presence of SARS-CoV-2 RNA. Results, expressed as cycle threshold will be then compared to analyze viral loads from the two different sites.

Moreover, an aliquot will be retro-transcribed into cDNA and sequenced by Next Generation Sequencing (NGS) to obtain the virus entire genome sequence or evaluated by RT-PCR for variant determination.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to IRCCS Sacro Cuore Don Calabria Hospital or health care workers or their family members. Among the family members, also children >4 years old will be included.
* Subjects verified as positive to SARS-CoV-2 according to either a molecular or antigen test, performed on nasopharyngeal swab, according to current diagnostics.
* Subjects who will accept to participate to the study and will sign the informed consent.

Exclusion Criteria:

* lack of any needed data or inform consent

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 real time RT-PCR analysis results of the nose and mouth swabs. | 2 months
  SARS-CoV-2 real time RT-PCR analysis results of the nose and mouth swabs.
- Droplet digital PCR (ddPCR) results for SARS-CoV-2 | 2 months
  - Droplet digital PCR (ddPCR) results for SARS-CoV-2
- NGS or RT-PCR results for genomic lineages or variant identification. | 2 months
  - NGS or RT-PCR results for genomic lineages or variant identification.
- RT-PCR analysis results for subgenomics | 2 months
  - RT-PCR analysis results for subgenomics

SECONDARY OUTCOMES:
SARS-CoV-2 real time RT-PCR analysis results of the nose and mouth swabs in relationship to the sampling site, to the viral characterization and to the time from diagnosis. | 2 months
  SARS-CoV-2 real time RT-PCR analysis results of the nose and mouth swabs in relationship to the sampling site, to the viral characterization and to the time from diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona, Italy